CLINICAL TRIAL: NCT02671136
Title: Hyperbaric Oxygen Therapy as Adjunctive Therapy to Scaling and Root-planing in the Management of Periodontitis in Patients With Type 2 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of subjects
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5150307
Record Dates: First submitted 2015-10-06; First posted 2016-02-02 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Diabetes; Periodontitis
MeSH Terms: conditions — Diabetes Mellitus; Periodontitis | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CWC with HBO (Other): Conventional Wound Therapies (CWC) with adjunctive Hyperbaric Oxygen Therapy
  Interventions: Device: Hyperbaric Oxygen therapy; Other: Conventional Wound Therapies
- CWC without HBO (Other): Conventional Wound Therapies (CWC) without adjunctive Hyperbaric Oxygen Therapy
  Interventions: Other: Conventional Wound Therapies

INTERVENTIONS:
Device: Hyperbaric Oxygen therapy
  Arms: CWC with HBO
Other: Conventional Wound Therapies

SUMMARY:
Diabetes and Periodontitis are both prevalent diseases affecting millions of Americans. Periodontitis is prevalent among Diabetics. Furthermore, Periodontitis and associated inflammation can increase insulin resistance in Diabetics and worsens the condition. Hyperbaric Oxygen Therapy (HBOT) has the potential to improve periodontal treatment outcome in poorly controlled diabetics. The study will compare periodontal treatment (SRP) outcome between 2 main diabetic type 2 patient groups receiving medical care treatment: either Conventional Wound Therapies (CWC) with or without adjunctive Hyperbaric Oxygen Therapy at LLU Health.

24 poorly controlled diabetic mellitus (DM) type 2 subjects (HbA1c =>7%) with Periodontitis will be assigned into the study arms HBO therapy and Non HBO therapy, based on their medical needs.

For all subjects demographic data (age, gender, ethnicity, smoking history, alcohol use history, BMI, current medication list) and oral health habits will be obtained. Blood samples for HbA1c determinations, clinical periodontal measurements (plaque index, probing measurements including pocket depth, attachment levels, gingival index and bleeding-on-probing) and subgingival microbial samples will be obtained at baseline and end of the study. Subgingival microbial samples will be collected from three randomly selected sites and analyzed for detection of about 300 of the most prevalent oral bacterial species. Differences in periodontal clinical outcomes and bacterial profiles will be identified utilizing ANCOVA (Analysis of Covariance).

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 2 (HbA1c =>7%)
* Generalized moderate to severe chronic periodontitis.
* Minimum of 10 permanent teeth
* Registered LLU patients

Exclusion Criteria:

* Well controlled Diabetes type 2
* Other systematic conditions with known associations to periodontitis
* Intra-oral conditions which may interfere with the accuracy of periodontal probing
* BMI greater than 45%

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Khocht, DDS, Principal Investigator — Faculty
Locations (1):
- Loma Linda University, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CWC With HBO: Conventional Wound Therapies (CWC) with adjunctive Hyperbaric Oxygen Therapy
  Hyperbaric Oxygen therapy
  Conventional Wound Therapies
- CWC Without HBO: Conventional Wound Therapies (CWC) without adjunctive Hyperbaric Oxygen Therapy
  Conventional Wound Therapies
Period: Overall Study
Arm/Group | CWC With HBO | CWC Without HBO
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This project was terminated early due to not enough subjects recruited.
Groups:
- Total: Total of all reporting groups
Arm/Group | CWC With HBO | CWC Without HBO | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Counts of Each Subgingival Bacterial Species
Description: Subgingival microbial samples will be obtained at baseline and end of the study. Subgingival microbial samples will be collected from three randomly selected sites with probing depth =>5mm. Collected microbial samples will be processed for HOMINGS analysis (The Human Oral Microbe Identification Microarray). Counts and proportions of each bacterial species will be determined for each subject and then averaged across subjects in the two groups. Differences in bacterial profiles will be analyzed using the repeated measures ANCOVA (Analysis of Covariance) procedure for paired observations.
Time Frame: 12 weeks
Population: No analysis conducted due to not enough subjects recruited and study terminated early.
Arm/Group | CWC With HBO | CWC Without HBO
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: No adverse event data collected. Study terminated early due to not enough subjects enrolled.
Description: No adverse event data collected. Study terminated early due to not enough subjects enrolled.
Arm/Group | CWC With HBO | CWC Without HBO
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT02671136/Prot_SAP_000.pdf